CLINICAL TRIAL: NCT00401154
Title: Pediatric Endurance and Limb Strengthening (PEDALS)
Brief Title: Study of a Stationary Cycling Intervention for Children With Spastic Diplegic Cerebral Palsy
Acronym: PEDALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Physical Therapy Clinical Research Network (Network)
Responsible Party: Principal Investigator, Sharon K. DeMuth, Assistant Professor of Clinical Physical Therapy, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HS-025023-CR001
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Spastic Diplegic Cerebral Palsy
Keywords: Spastic Diplegia; Cerebral Palsy; Children; Adolescents; Strengthening; Endurance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Stationary Cycling (Experimental): Subjects receiving the intervention performed stationary cycling 3 times a week for 30 sessions over 12 weeks.
  Interventions: Other: Stationary Cycling

INTERVENTIONS:
Other: Stationary Cycling — Use of a stationary bicycle for exercise

SUMMARY:
The study is about the effect of an exercise program using stationary bicycling for children with the spastic diplegic form of cerebral palsy. Spastic diplegia is a type of cerebral palsy that involves spasticity or "tightness" of the leg muscles. We hope to learn whether this type of exercise will allow the children to develop improved strength in the muscles that bend and straighten their knees, enhance their level of physical fitness, improve their ability to walk and improve their ability to perform other activities that are important to them. We hypothesize that children who participate in the stationary cycling intervention will gain strength in the muscles that bend and straighten their knees, will be able to complete a 600 yard walk run test (a test of endurance) more rapidly, and will improve their score on a test of function called the Gross Motor Function Measure (a test designed specifically for children with cerebral palsy).

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 7 and 16 years and engaged in regular education as their primary academic path (children receiving resource help will not be excluded); - ability to follow simple verbal directions;
* good or fair selective motor control for at least one limb; and
* ability to walk independently, with or without assistive devices, for short distances. The lowest level of walking ability for inclusion is independent walking indoors but limitations outdoors and in the community, requiring the use of a wheelchair in these settings. These criteria for walking ability place subjects in Levels I-III of the Gross Motor Functional Classification System (GMFCS) (Palisano et al., 1997).

Exclusion Criteria:

* musculoskeletal or neurosurgical surgery or baclofen pump implantation within the past year;
* botulinum toxin injections within the past 6 months;
* serial casting or new orthotics within the past 3 months;
* initiating or increasing oral medications that affect the neuromuscular system, e.g. baclofen, within the past 3 months;
* onset of physical therapy, exercise, sport activity, or change in assistive devices for walking within the past 3 months;
* inability or unwillingness to maintain age appropriate behavior;
* serious medical conditions such as cardiac disease, diabetes, asthma, or uncontrolled seizures;
* current participation in a fitness program, that includes a cardiorespiratory endurance exercise, at least one time per week;
* significant hip joint contractures so that the hip cannot be passively moved throughout an excursion between 30 and 80 degrees;
* significant knee joint contractures so that the knee cannot be passively moved throughout an excursion between 40 and 110 degrees; and
* significant ankle joint contractures so that the ankle cannot be passively moved throughout an excursion of -10 to 20 degrees of plantarflexion. Exclusion criteria 8 - 10 are based on passive joint excursions necessary to perform stationary cycling (Ericson et al., 1988) allowing for some hip and knee joint compensation for subjects without ankle dorsiflexion range of motion.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2003-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-66 (GMFM) | Basline and Post Intervention
  Describes gross motor function in children with cerebral palsy.
600 Yard Walk-Run Test | Baseline and Post Intervention
  Timed test to show how rapidly the subject can walk or run 600 yards.
30 Second Walk Test | Basline and Post Intervention
  Timed test to measure the distance a subject walks in 30 seconds.
Knee Flexor and Knee Extensor Torque | Basline and Post Intervention
  Measures strength of the knee flexors and extensor muscles.
Pediatric Quality of Life Inventory (PedsQL) | Basline and Post Intervention
  Questionnaire that assesses quality of life
Pediatric Outcomes Data Collection Instrument (PODCI) | Basline and Post Intervention
  Questionnaire that assesses health related quality of life

SECONDARY OUTCOMES:
Gait Analysis will be performed on a subset of the children enrolled. | Basline and Post Intervention
  Analyses changes in walking

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Fowler, PT, PhD, Principal Investigator — University of California at Los Angeles
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Demuth SK, Knutson LM, Fowler EG. The PEDALS stationary cycling intervention and health-related quality of life in children with cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2012 Jul;54(7):654-61. doi: 10.1111/j.1469-8749.2012.04321.x. Epub 2012 May 14. PMID 22582760
- [Derived] Fowler EG, Knutson LM, Demuth SK, Siebert KL, Simms VD, Sugi MH, Souza RB, Karim R, Azen SP; Physical Therapy Clinical Research Network (PTClinResNet). Pediatric endurance and limb strengthening (PEDALS) for children with cerebral palsy using stationary cycling: a randomized controlled trial. Phys Ther. 2010 Mar;90(3):367-81. doi: 10.2522/ptj.20080364. Epub 2010 Jan 21. PMID 20093327